CLINICAL TRIAL: NCT07174193
Title: Piezosurgery Versus Conventional Techniques in Orthognathic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Tim Knuppe, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PiezoOrthognathicSurgery
Record Dates: First submitted 2025-08-10; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Orthognathic Surgical Procedures; Piezoelectric Technique
Keywords: orthognathic surgery; piezosurgery
MeSH Terms: interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezosurgery (Experimental): Patients undergoing BSSO with piezosurgery
  Interventions: Device: Piezosurgery
- Conventional group (Active Comparator): Patients undergoing BSSO with conventional techniques
  Interventions: Device: Conventional techniques

INTERVENTIONS:
Device: Piezosurgery — Initially introduced in the field of implantology, piezosurgery has gained increasing popularity in orthognathic surgery in recent years (7-9). This technique utilizes ultrasonic vibrations ranging from 60-210 μm/s at frequencies between 24-29 kHz to cut bone, thereby minimizing trauma to surrounding soft tissue (10). Although numerous studies have been conducted, many clinical investigations have been limited by small sample sizes and insufficiently described methodologies (17, 18). Furthermore, the lack of standardized assessment tools hinders reliable comparisons of outcomes across studies (19). While surgeons increasingly recommend the use of piezosurqical instruments in orthognathic surgery, robust evidence from the literature remains insufficient to support the change in surgical technique.
  Arms: Piezosurgery
Device: Conventional techniques — In the control group a Lindemann burr will be used to perform the horizontal and vertical osteotomies and the cut at the lower border of the mandible. A reciprocal saw will then be used to connect the horizontal and vertical osteotomies in the sagittal plane.
  Arms: Conventional group

SUMMARY:
The goal of this randomized double-blinded controlled clinical trial is to determine whether piezosurgery can reduce complications and improve outcomes compared to conventional osteotomy techniques in patients undergoing bilateral sagittal split osteotomy (BSSO), with or without concurrent Le Fort I osteotomy (bimaxillary surgery).

The main questions this study aims to answer are:

* Does piezosurgery reduce inferior alveolar nerve impairment following BSSO compared to conventional techniques?
* Does piezosurgery affect surgical duration, intraoperative blood loss, rates of bad splits, postoperative infections, costs, and environmental sustainability compared to conventional techniques?

Researchers will compare BSSO performed with piezosurgery versus BSSO performed with conventional oscillating saw and burr techniques to see if piezosurgery leads to better sensory outcomes, reduced morbidity, and improved cost-effectiveness and sustainability.

Participants will be:

* Dutch or English-speaking adults aged 18-65 scheduled for BSSO or BIMAX surgery at Erasmus Medical Centre (Rotterdam) or St. Anna Hospital (Geldrop, Netherlands).
* Exclusions include bone healing disorders, coagulation issues, facial trauma history, smoking, craniofacial anomalies, and planned simultaneous genioplasty.

Participants will:

* Undergo preoperative assessment of inferior alveolar nerve function (two-point discrimination test, validated questionnaire).
* Be randomized into:

  * Intervention group: BSSO performed entirely using piezosurgery.
  * Control group: BSSO performed with conventional burr and saw techniques.
* Have their surgery performed by experienced maxillofacial surgeons following standardized protocols.
* Have operative time and blood loss recorded during surgery.
* Be followed up at 1 week, 3 months, 6 months, and 1 year for nerve function, sensory recovery, and infection assessment.
* Complete postoperative questionnaires on sensory changes at 3 months and 1 year.
* Have surgical outcomes evaluated by blinded examiners.
* Contribute to a life cycle cost analysis (LCC) and life cycle assessment (LCA) comparing equipment cost, maintenance, energy use, waste generation, and environmental impact between techniques.

DETAILED DESCRIPTION:
This is a randomized, double-blinded controlled clinical trial designed to evaluate the efficacy, safety, cost-effectiveness, and environmental impact of piezosurgery compared to conventional osteotomy techniques in orthognathic surgery. The study focuses on patients undergoing bilateral sagittal split osteotomy (BSSO), either as a standalone procedure or combined with Le Fort I osteotomy (bimaxillary surgery).

Orthognathic surgery is a well-established treatment for dentofacial deformities, performed to correct occlusal discrepancies and improve both function and aesthetics. The conventional technique for mandibular osteotomy employs rotary and oscillating instruments, which may increase the risk of iatrogenic injury to the inferior alveolar nerve, intraoperative bleeding, and postoperative swelling. Piezosurgery, a technique utilizing ultrasonic microvibrations for selective bone cutting, has been proposed to minimize trauma to adjacent soft tissues, potentially reducing sensory deficits and improving recovery.

Study Rationale Preliminary evidence from smaller clinical studies suggests that piezosurgery may lower the incidence of inferior alveolar nerve impairment, reduce intraoperative bleeding, and lessen postoperative morbidity, but it may also increase operative time. Many prior studies have been limited by small sample sizes, heterogeneous methodologies, and lack of standardized neurosensory assessment. This trial addresses these limitations with adequate statistical power, standardized testing, and rigorous blinding procedures.

Intervention and Control

Intervention arm: All osteotomy cuts performed using piezosurgical devices.

Control arm: Osteotomy performed using a Lindemann burr for horizontal and vertical cuts, followed by a reciprocating saw to connect osteotomies.

The allocation ratio is 1:1, determined via block randomization in Castor EDC with variable block sizes (2, 4, and 6).

Blinding Participants will remain blinded to treatment allocation. Postoperative neurosensory assessments will be conducted by independent examiners blinded to group assignment.

Procedures All participants will undergo standardized preoperative assessment of inferior alveolar nerve function, including the static two-point discrimination test and a validated questionnaire on subjective sensory changes. Surgeries will be performed by experienced maxillofacial surgeons using the Hunsuck modification of the BSSO technique.

Intraoperative metrics will include surgical duration (from incision to final suture) and quantified blood loss (suction volume minus irrigation fluid plus gauze weight). Adverse intraoperative events such as "bad splits" will be documented. Postoperative infection will be defined according to CDC criteria.

Follow-up will occur at 1 week, 3 months, 6 months, and 12 months postoperatively. Neurosensory function will be reassessed at each visit, and the validated patient questionnaire will be completed at 3 months and 12 months.

Cost and Sustainability Assessment A life cycle cost analysis (LCC) will compare acquisition, operation, maintenance, and disposal costs between the two techniques. A life cycle assessment (LCA) will evaluate environmental impact, including CO₂ emissions, energy consumption, sterilization requirements, and waste generation.

Sample Size Sample size calculations were based on detecting clinically meaningful differences in operative time, blood loss, and nerve injury rates. The largest required sample size was 31 participants per group to detect differences in nerve impairment at 3-6 months with 80% power and α = 0.05.

Statistical Analysis Primary outcome (time to functional sensory recovery) will be analyzed using Kaplan-Meier survival curves and the log-rank test. Neurosensory scores will be compared using Chi-square or Fisher's exact tests. Continuous secondary outcomes will be analyzed using Student's t-test or Mann-Whitney U test depending on distribution. Categorical outcomes (e.g., bad split, infection) will be compared using Chi-square or Fisher's exact tests. The relationship between surgeon experience with piezosurgery and operative time will be explored using linear regression. A p-value < 0.05 will be considered statistically significant.

This trial is designed to provide robust evidence regarding both clinical and economic implications of adopting piezosurgery in orthognathic surgery.

ELIGIBILITY:
4.2 Inclusion criteria

We will include:

* Dutch or English-speaking patients
* Patients 18-65 years of age

4.3 Exclusion criteria

The following patients will be excluded from the study:

* Patients with any underlying comorbidities or medication use that may impair bone healing, i.e., radiotherapy in the head- and neck region or the use of antiresorptive drugs.
* Patients with coagulation disorders or those using of anticoagulative medication
* Patients with a history of facial trauma or previous facial surgery
* Patients who smoke
* Patients with facial cleft(s) or other craniofacial anomalies
* Patients undergoing simultaneous genioplasty

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Inferior alveolar nerve impairment following BSSO measured using the static two-point discrimination test (Weber test). Functional recovery will be evaluated using the sensory evaluation scale. | Measurements will be done 1 week post-op, 3 months post-op, 6 months post-op and 1 year post-op.
  Inferior alveolar nerve impairment will be assessed using the static two-point discrimination test (Weber test). The procedure will first be explained and demonstrated on the patients' hands to ensure comprehension. Testing will take place in a quiet room, with the patient seated and the eyes closed. A blinded examiner will perform the Weber test using a two-point discriminator to stimulate predetermined facial areas. Patients will be instructed to indicate whether they perceive one or two distinct points. To minimize variability due to inconsistent stimulus pressure, flexible calibrated filaments will be used. The reliability of neurosensory assessment will be reinforced by applying the staircase method, as described by Van der Cruysse et al.

SECONDARY OUTCOMES:
To evaluate the impact of piezosurgery on surgical duration in orthognathic procedures compared to conventional techniques. | Data will be gathered during surgery.
  Operative time will be defined as the duration (in minutes) from the initial incision to the final suture.
To assess intraoperative blood loss associated with piezosurgery versus conventional techniques in orthognathic procedures. | Data will be gathered during surgery.
  Intraoperative blood loss will be quantified by measuring the volume (in mL) collected via suction, subtracting the amount of surgical rinsing and cooling fluid. Only intraoperative blood loss during a BSSO procedures will be considered to avoid result distortion from maxillary blood loss in BIMAX cases.
To examine the incidence of postoperative infections following orthognathic procedures using piezosurgery compared to conventional techniques. | Assessments will be done up to 1 year after surgery.
  Surgical site infection (SSI) will be defined according to the criteria outlined by the Centers for Disease Control and Prevention (CDC). An SSI is diagnosed when osteosynthesis material is used and an infection occurs within one year postoperatively. Infections are identified by the presence of clinical symptoms and the need for antibiotic treatment.
To compare the incidence of bad splits during BSSO between piezosurgery and conventional techniques. | Data will be gathered during surgery.
  Bad split is defined as an unfavorable and and unanticipated split pattern of the mandible that requires additional fixation techniques or may lead to the termination of the procedure.
To analyze the costs associated with use of piezosurgery versus conventional techniques in orthognathic procedures using a life cycle costing model. | Data will be gathered one year after start of inclusion.
  Cost comparison between piezosurgery and conventional techniques will be performed using a life cycle costing (LCC). This analysis will include purchasing costs, device lifetime, cleaning costs, maintenance costs and waste disposal costs (26).
To investigate the sustainability of piezosurgery in comparison with conventional techniques in orthognathic procedures using a life cylce assessment. | Data will be gathered one year after start of inclusion.
  Life cycle assessment (LCA) will be used to evaluate the environmental impact of piezosurgery versus conventional techniques. LCA accounts for direct emissions during product use, as well as emissions during manufacturing and disposal processses (27).
To investigate the influence of surgical experience with piezosurgery on procedure duration in orthognathic procedures. | Information will be gathered during surgery.
  Surgeon experience will be quantified by the number of osteotomies performed using piezosurgery. None of the participating surgeons routinely used piezosurgery in orthognathic surgery using piezosurgery prior to the start of this study.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Anna Ziekenhuis, Geldrop
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided